CLINICAL TRIAL: NCT02907216
Title: Immunogenicity and Safety of the Diphtheria, Tetanus, Pertussis and Inactivated Poliovirus (DPT-IPV) Vaccine Squarekids Co-administered With GSK Biologicals' Human Rotavirus (HRV) Vaccine Rotarix (GSK444563) in Healthy Infants
Brief Title: Evaluation of Immunogenicity and Safety of the Diphtheria, Tetanus, Pertussis and Inactivated Poliovirus (DPT-IPV) Vaccine Squarekids Co-administered With GSK Biologicals' Human Rotavirus (HRV) Vaccine Rotarix (GSK444563) in Healthy Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114720; 2014-005282-78 (EudraCT Number)
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Rotavirus
Keywords: Healthy Japanese infants; Safety; Diphtheria, Tetanus, Pertussis and Inactivated Poliovirus (DPT-IPV) vaccine; Vaccination; Oral HRV liquid vaccine; Immunogenicity
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — RIX4414 vaccine

ARMS (2):
- Co-administration Group (Experimental): Subjects aged 6 to 12 weeks who receive the Squarekids vaccine (diphtheria, tetanus, pertussis and inactivated poliovirus [DPT-IPV] vaccine) according to a 3, 4, 6 month schedule and the liquid Rotarix vaccine (oral live attenuated human rotavirus [HRV] vaccine) according to a 2, 3 month schedule. The HRV vaccine is administered orally while the DTP-IPV vaccine is administered subcutaneously in the upper arm or upper thigh.
  Interventions: Biological: Squarekids; Biological: Rotarix
- Staggered Group (Active Comparator): Subjects aged 6 to 12 weeks who receive the Squarekids vaccine (diphtheria, tetanus, pertussis and inactivated poliovirus [DPT-IPV] vaccine) according to a 3, 4.5, 6 month schedule and the liquid Rotarix vaccine (oral live attenuated human rotavirus [HRV] vaccine) according to a 2, 3.5 month schedule. The HRV vaccine is administered orally while the DTP-IPV vaccine is administered subcutaneously in the upper arm or upper thigh.
  Interventions: Biological: Squarekids; Biological: Rotarix

INTERVENTIONS:
Biological: Squarekids — Three doses administered subcutaneously in the upper arm or thigh
Biological: Rotarix — Two doses administered orally

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the diphtheria, tetanus, pertussis and inactivated poliovirus (DPT-IPV) vaccine Squarekids administered with or without the GSK Biologicals' liquid Rotarix (HRV) vaccine, in healthy Japanese infants aged 6 - 12 weeks. GSK Biologicals' liquid HRV vaccine Rotarix is licensed in Japan since 2011. Although the concomitant administration of GSK Biologicals' DTP-IPV vaccine has been evaluated during the clinical development of the HRV vaccine, the vaccine differed in composition and route of administration from the DPT-IPV vaccine Squarekids manufactured in Japan. Hence, as requested by the Japanese regulatory authorities, this post-licensure study will evaluate the immunogenicity of the DPT-IPV vaccine manufactured in Japan when co-administered with the liquid HRV vaccine

DETAILED DESCRIPTION:
This study is a phase IV, open-label, randomised, controlled, multi-centric, single-country study with two parallel groups. Subjects in the co-administration group will be administered the DPT-IPV vaccine according to a 3, 4, 6 month schedule and the liquid HRV vaccine according to a 2, 3 month schedule. Subjects in the staggered group will be administered the DPT-IPV vaccine according to a 3, 4.5, 6 month schedule and the liquid HRV vaccine according to a 2, 3.5 month schedule. The intended duration of the study, per subject, is 5 months.

A sub-cohort of subjects (HRV Immunogenicity sub-cohort) from both the study groups will include the first 73 subjects enrolled into the study to assess the serum anti-RV IgA seropositivity and Geometric Mean Concentrations (GMC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/ Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first dose of HRV vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term as per the delivery records.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days before the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone (≥ 0.5 mg/kg/day, or equivalent). Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not fore-seen by the study protocol within the period starting 30 days before the first dose of HRV vaccine administration and ending at Visit 7, with the exception of other routinely administered vaccines like PCV, Hib, BCG, hepatitis B, meningococcal vaccine and inactivated influenza vaccines, which are allowed at any time during the study, if administered at sites different from the sites used to administer the DPT-IPV vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Uncorrected congenital malformation of the gastrointestinal tract that would predispose for Intussusception (IS).
* History of IS.
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* Previous vaccination against rotavirus, diphtheria, tetanus, pertussis and/ or poliovirus.
* Previous confirmed occurrence of RV GE, diphtheria, tetanus, pertussis, and/ or polio disease.
* GE within 7 days preceding the HRV vaccine administration.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the HRV or DPT-IPV vaccines.
* Hypersensitivity to latex.
* History of any neurological disorders or seizures.
* History of SCID.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F on oral, axillary or tympanic setting, or ≥ 38.0°C /100.4°F on rectal setting.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 292 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19839

REFERENCES:
- [Background] Gillard P, Tamura T, Kuroki H, Morikawa Y, Moerman L, Parra J, Kitamura Y, Mihara K, Okamasa A. Immunogenicity and safety of the diphtheria, pertussis, tetanus and inactivated poliovirus vaccine when co-administered with the human rotavirus vaccine (Rotarix) in healthy Japanese infants: a phase IV randomized study. Hum Vaccin Immunother. 2019;15(4):800-808. doi: 10.1080/21645515.2018.1564441. Epub 2019 Feb 20. PMID 30785851

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 292 subjects enrolled in the study, the first 73 subjects enrolled into each of the 2 study groups (total of 146 subjects) were allocated to the HRV immunogenicity sub-cohort to evaluate immunogenicity of the liquid HRV vaccine.
Groups:
- Co-administration Group: Subjects aged 6 to 12 weeks who received the Squarekids vaccine (diphtheria, tetanus, pertussis and inactivated poliovirus [DPT-IPV] vaccine) according to a 3, 4, 6 month schedule and the liquid Rotarix vaccine (oral live attenuated human rotavirus [HRV] vaccine) according to a 2, 3 month schedule. The HRV vaccine was administered orally while the DTP-IPV vaccine was administered subcutaneously in the upper arm or upper thigh.
- Staggered Group: Subjects aged 6 to 12 weeks who received the Squarekids vaccine (diphtheria, tetanus, pertussis and inactivated poliovirus [DPT-IPV] vaccine) according to a 3, 4.5, 6 month schedule and the liquid Rotarix vaccine (oral live attenuated human rotavirus [HRV] vaccine) according to a 2, 3.5 month schedule. The HRV vaccine was administered orally while the DTP-IPV vaccine was administered subcutaneously in the upper arm or upper thigh.
Period: Overall Study
Arm/Group | Co-administration Group | Staggered Group
Started | 147 | 145
Completed | 146 | 144
Not Completed | 1 | 1
Not completed — No benefit to be obtained by continuing | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Co-administration Group: Subjects aged 6 to 12 weeks who received the DPT-IPV vaccine according to a 3, 4, 6 month schedule and the liquid HRV vaccine according to a 2, 3 month schedule. The HRV vaccine was administered orally while the DTP-IPV vaccine was administered subcutaneously in the upper arm or upper thigh.
- Staggered Group: Subjects aged 6 to 12 weeks who received the DPT-IPV vaccine according to a 3, 4.5, 6 month schedule and the liquid HRV vaccine according to a 2, 3.5 month schedule. The HRV vaccine was administered orally while the DTP-IPV vaccine was administered subcutaneously in the upper arm or upper thigh.
- Total: Total of all reporting groups
Arm/Group | Co-administration Group | Staggered Group | Total
Number analyzed (Participants) | 147 | 145 | 292
Age, Continuous [Mean (Standard Deviation); unit: Weeks]
  Weeks of age at Dose 1 of HRV | 9.5 (1.1) | 9.4 (1.1) | 9.5 (1.1)
  Weeks of age at Dose 2 of HRV | 14 (1.1) | 15.5 (1.3) | 14.7 (1.4)
  Weeks of age at Dose 1 of DPT-IPV | 14 (1.1) | 13.9 (1) | 14 (1.1)
  Weeks of age at Dose 2 of DPT-IPV | 18.5 (1.2) | 20 (1.4) | 19.2 (1.5)
  Weeks of age at Dose 3 of DPT-IPV | 23.7 (1.8) | 25 (1.9) | 24.4 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 65 | 137
  Male | 75 | 80 | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese Heritage | 147 | 145 | 292

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations Greater Than or Equal to (≥) the Cut-off Value
Description: Percentage of subjects with anti-D and anti-T antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: One month post third dose of DTP-IPV vaccine (At Month 5)
Population: Analysis was performed on According-to-Protocol (ATP) cohort which included all subjects who complied with vaccination schedules of DPT-IPV and HRV vaccines, complied with the blood sampling schedule and for whom immunogenicity data was available for at least for one antigen of the DPT-IPV vaccine at Visit 7 (Month 5) sampling time point.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 141 | 138
Percentage of subjects
  Anti-D antibody ≥ 0.1 IU/mL: number analyzed (Participants) | 141 | 137
  Anti-D antibody ≥ 0.1 IU/mL | 100 [97.4 to 100] | 100 [97.3 to 100]
  Anti-T antibody ≥ 0.1 IU/mL | 98.6 [95 to 99.8] | 99.3 [96 to 100]
Statistical Analysis 1: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-D antibody concentration ≥ 0.1 IU/mL; Test type: Non-Inferiority — Criteria for non-inferiority: The Lower Limit (LL) of the standardised asymptotic 95% Confidence Interval (CI) on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective concentrations ≥ 0.1 IU/mL for anti-D antibodies should be ≥ -10%; Difference-Seroprotective concentration = 0, 95% CI 2-sided [-2.66 to 2.74] — The 2-sided asymptotic standardised 95% CIs for the difference between groups in terms of percentage of subjects with antibody concentration ≥ to the pre-defined cut-off
Statistical Analysis 2: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-T antibody concentration ≥ 0.1 IU/mL; Test type: Non-Inferiority — Criteria for non-inferiority: The LL of the standardised asymptotic 95% CI on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective concentrations ≥ 0.1 IU/mL for anti-T antibodies should be ≥ -10%; Difference-Seroprotective concentration = -0.69, 95% CI 2-sided [-4.39 to 2.71] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Subjects With Anti-pertussis Toxoid (Anti-PT) and Anti-filamentous Haemagglutinin (Anti-FHA) Antibody Concentrations ≥ the Cut-off Value
Description: Percentage of subjects with anti-PT and anti-FHA antibody concentrations ≥ 10 IU/mL.
Time Frame: One month post third dose of DTP-IPV vaccine (At Month 5)
Population: Analysis was performed on ATP cohort which included all subjects who complied with vaccination schedules of DPT-IPV and HRV vaccines, complied with the blood sampling schedule and for whom immunogenicity data was available for at least for one antigen of the DPT-IPV vaccine at Visit 7 (Month 5) sampling time point.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 141 | 138
Percentage of subjects
  Anti-PT antibody ≥ 10 IU/mL | 95.7 [91 to 98.4] | 92.8 [87.1 to 96.5]
  Anti-FHA antibody ≥ 10 IU/mL | 100 [97.4 to 100] | 100 [97.4 to 100]
Statistical Analysis 1: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-PT antibody concentration ≥ 10 IU/mL; Test type: Non-Inferiority — Criteria for non-inferiority: The LL of the standardised asymptotic 95% CI on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective concentrations ≥ 10 IU/mL for anti-PT antibodies should be ≥ -10%; Difference-Seroprotective concentration = 2.99, 95% CI 2-sided [-2.7 to 9.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-FHA antibody concentration ≥ 10 IU/mL; Test type: Non-Inferiority — Criteria for non-inferiority: The LL of the standardised asymptotic 95% CI on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective concentrations ≥ 10 IU/mL for anti-FHA antibodies should be ≥ -10%; Difference-Seroprotective concentration = 0, 95% CI 2-sided [-2.66 to 2.72] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Percentage of Subjects With Anti-poliovirus Serotypes 1, 2 and 3 (Anti-polio 1, 2 and 3) Antibody Titers ≥ the Cut-off Value
Description: Percentage of subjects with anti-polio 1, 2 and 3 antibody titers ≥ 8 estimated doses 50% (ED50).
Time Frame: One month post third dose of DTP-IPV vaccine (At Month 5)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 140 | 137
Percentage of subjects
  Anti-Polio 1 antibody ≥ 8 ED50 | 100 [97.4 to 100] | 100 [97.3 to 100]
  Anti-Polio 2 antibody ≥ 8 ED50: number analyzed (Participants) | 128 | 127
  Anti-Polio 2 antibody ≥ 8 ED50 | 100 [97.2 to 100] | 100 [97.1 to 100]
  Anti-Polio 3 antibody ≥ 8 ED50: number analyzed (Participants) | 132 | 123
  Anti-Polio 3 antibody ≥ 8 ED50 | 100 [97.2 to 100] | 99.2 [95.6 to 100]
Statistical Analysis 1: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-polio 1 seroprotective titres ≥ 8 ED50; Test type: Non-Inferiority — Criteria for non-inferiority: The LL of the standardised asymptotic 95% CI on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective titers ≥ 8 ED50 for anti-polio 1 antibodies should be ≥ -10%; Difference in seroprotective titer = 0, 95% CI 2-sided [-2.68 to 2.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-polio 2 seroprotective titres ≥ 8 ED50; Test type: Non-Inferiority — Criteria for non-inferiority: The LL of the standardised asymptotic 95% CI on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective titers ≥ 8 ED50 for anti-polio 2 antibodies should be ≥ -10%; Difference in seroprotective titer = 0, 95% CI 2-sided [-2.92 to 2.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Co-administration Group vs Staggered Group; Difference between Co-administration Group minus Staggered Group in terms of percentage of subjects with anti-polio 3 seroprotective titres ≥ 8 ED50; Test type: Non-Inferiority — Criteria for non-inferiority: The LL of the standardised asymptotic 95% CI on the difference (Co-administration Group minus Staggered Group) in the percentage of subjects with seroprotective titers ≥ 8 ED50 for anti-polio 3 antibodies should be ≥ -10%; Difference in seroprotective titer = 0.81, 95% CI 2-sided [-2.04 to 4.47] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Seropositive Subjects for Serum Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibodies in a Sub-cohort of Subjects
Description: A seropositive subject for serum anti-RV IgA antibodies was defined as a subject with anti-RV IgA antibody concentration ≥ the seropositivity cut-off value of 20 units per milliliter (U/mL). Immunogenicity of the liquid HRV vaccine in terms of serum anti-RV IgA antibody seropositivity was assessed in a sub-cohort of subjects (HRV immunogenicity sub-cohort) which included the first 73 subjects enrolled into each of the 2 study groups.
Time Frame: One month post second dose of liquid HRV vaccine (At Month 2 for the Co-administration Group and at Month 2.5 for the Staggered Group)
Population: Analysis was performed on HRV immunogenicity sub-cohort of ATP cohort which included all subjects who complied with vaccination schedules of DPT-IPV and HRV vaccines, complied with the blood sampling schedule and for whom immunogenicity data was available for at least for one antigen of the DPT-IPV vaccine at Visit 7 (Month 5) sampling time point.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 69 | 67
Percentage of subjects | 92.8 [83.9 to 97.6] | 92.5 [83.4 to 97.5]

5. Secondary Outcome: Serum Anti-RV IgA Antibody Concentration to Evaluate Immunogenicity in a Sub-cohort of Subjects
Description: Concentration of serum anti-RV IgA antibody was assessed by Enzyme Linked Immunosorbent Assay (ELISA) and expressed as geometric mean concentration (GMC) in U/mL. The assay cut-off was 20 U/mL. Immunogenicity of the liquid HRV vaccine in terms of serum anti-RV IgA antibody GMC was assessed in a sub-cohort of subjects (HRV immunogenicity sub-cohort) which included the first 73 subjects enrolled into each of the 2 study groups.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 69 | 67
U/mL | 350.1 [223.3 to 548.8] | 362.5 [251 to 523.5]

6. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations to Evaluate Immunogenicity
Description: Concentrations of anti-D and anti-T antibodies were assessed by ELISA, presented as GMCs and expressed in IU/mL. The assay cut-off for anti-D and anti-T antibody concentrations was 0.1 IU/mL.
Time Frame: One month post third dose of DTP-IPV vaccine (At Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 141 | 138
IU/mL
  Anti-D antibody: number analyzed (Participants) | 141 | 137
  Anti-D antibody | 5.4 [4.9 to 6] | 6 [5.5 to 6.6]
  Anti-T antibody | 1.6 [1.3 to 2] | 2 [1.7 to 2.4]

7. Secondary Outcome: Anti-polio 1, 2 and 3 Antibodies Titers to Evaluate Immunogenicity
Description: Titers of anti-polio 1, 2 and 3 were assessed by Neutralisation Assay (NEU) and presented as Geometric Mean Titers (GMTs). The assay cut-off was 8 ED50.
Time Frame: One month post third dose of DTP-IPV vaccine (At Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 140 | 137
Titer
  Anti-Polio 1 antibody | 404.7 [341.4 to 479.8] | 427.9 [359.3 to 509.6]
  Anti-Polio 2 antibody: number analyzed (Participants) | 128 | 127
  Anti-Polio 2 antibody | 371 [307 to 448.5] | 470.6 [388.3 to 570.3]
  Anti-Polio 3 antibody: number analyzed (Participants) | 132 | 123
  Anti-Polio 3 antibody | 436.3 [365.6 to 520.7] | 409.8 [330.8 to 507.5]

8. Secondary Outcome: Anti-PT and Anti-FHA Antibody Concentrations to Evaluate Immunogenicity
Description: Concentrations of anti-PT and anti-FHA antibodies were assessed by ELISA, presented as GMCs and expressed in IU/mL. The assay cut-offs for anti-PT and anti-FHA antibody concentrations were 2.693 IU/mL and 2.046 IU/mL respectively.
Time Frame: One month post third dose of DTP-IPV vaccine (At Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 141 | 138
IU/mL
  Anti-PT antibody | 31.5 [28.4 to 34.9] | 31.5 [27.9 to 35.6]
  Anti-FHA antibody | 83.7 [74.8 to 93.6] | 97.2 [86.7 to 109]

9. Secondary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs) After Each Dose of Liquid HRV Vaccine
Description: Assessed solicited general AEs were fever (defined as axillary temperature ≥ 37.5 degrees Celsius [°C]), irritability/fussiness, diarrhoea (defined as passage of three or more looser than normal stools within a day), vomiting (defined as one or more episodes of forceful emptying of partially digested stomach contents ≥ 1 hour after feeding within a day), loss of appetite and cough/runny nose. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 8-day (Days 0-7) follow-up period after each dose of liquid HRV vaccine
Population: Analysis was performed on the Total Vaccinated cohort (TVC) which included all subjects with at least one dose of the study vaccines administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 147 | 145
Participants
  Any Fever, Dose 1 | 31 | 32
  Any Irritability / Fussiness, Dose 1 | 66 | 62
  Any Diarrhoea, Dose 1 | 30 | 32
  Any Vomiting, Dose 1 | 19 | 19
  Any Loss of Appetite, Dose 1 | 18 | 10
  Any Cough, Dose 1 | 41 | 40
  Any Fever, Dose 2 | 31 | 15
  Any Irritability / Fussiness, Dose 2 | 61 | 41
  Any Diarrhoea, Dose 2 | 22 | 26
  Any Vomiting, Dose 2 | 14 | 18
  Any Loss of Appetite, Dose 2 | 17 | 9
  Any Cough, Dose 2 | 53 | 45

10. Secondary Outcome: Number of Subjects With Any Solicited Local AEs After First Dose of DTP-IPV Vaccine
Description: Assessed solicited local AEs were pain, redness and swelling at injection site. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 8-day (Days 0-7) follow-up period after first dose of DTP-IPV vaccine
Population: Analysis was performed on the TVC which included all subjects with at least one dose of the study vaccines administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 147 | 144
Participants
  Any Pain | 32 | 24
  Any Redness (mm) | 85 | 84
  Any Swelling (mm) | 50 | 44

11. Secondary Outcome: Number of Subjects With Any Solicited General AEs After First Dose of DTP-IPV Vaccine
Description: Assessed solicited general AEs were drowsiness, fever (defined as axillary temperature ≥ 37.5 °C), irritability/fussiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 8-day (Days 0-7) follow-up period after first dose of DTP-IPV vaccine
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 147 | 144
Participants
  Any Drowiness | 37 | 39
  Any Fever | 31 | 32
  Any Irritability / Fussiness | 61 | 59
  Any Loss of Appetite | 17 | 18

12. Secondary Outcome: Number of Subjects With Any Unsolicited AEs After Each Dose of Liquid HRV Vaccine
Description: Unsolicited AEs were defined as any AE reported in addition to those solicited during the clinical study and any solicited AE with onset outside the specified period of follow-up for solicited AEs. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after each dose of liquid HRV vaccine
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 147 | 145
Participants | 88 | 81

13. Secondary Outcome: Number of Subjects With Any Unsolicited AE After First Dose of DTP-IPV Vaccine
Description: as for outcome 12
Time Frame: During the 31-day (Days 0-30) follow-up period after first dose of DTP-IPV vaccine
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 147 | 144
Participants | 65 | 59

14. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Assessed SAEs included any untoward medical occurrence that resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (from Day 0 to Month 5)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Staggered Group
Number analyzed (Participants) | 147 | 145
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Solicited local & general AEs were reported during the 8-day (Days 0-7) post-vaccination period following first dose of DTP-IPV vaccine; solicited general AEs were reported during the 8-day (Days 0-7) post-vaccination period following each dose of liquid HRV vaccine. Unsolicited AEs were reported the 31-day (Days 0-30) post-vaccination period after the first dose of DTP-IPV vaccine & after each dose of liquid HRV vaccine. SAEs were reported during the entire study period (from Day 0 to Month 5).
Arm/Group | Co-administration Group | Staggered Group
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/145
Serious Adverse Events (participants affected / at risk) | 4/147 | 5/147
Other Adverse Events (participants affected / at risk) | 141/147 | 143/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administration Group (N=147) | Staggered Group (N=147)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administration Group (N=147) | Staggered Group (N=145)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 69 (95) | 72 (85)
Decreased appetite (Metabolism and nutrition disorders) | 27 (35) | 31 (37)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 41 (52) | 50 (61)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (10)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0)
Eczema infantile (Skin and subcutaneous tissue disorders) | 13 (14) | 11 (11)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 3 (3) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 85 (85) | 84 (84)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 32 (32) | 24 (24)
Injection site swelling (General disorders) | 50 (50) | 44 (44)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability postvaccinal (General disorders) | 93 (127) | 99 (162)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Leukoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 22 (26) | 33 (37)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (2)
Pyrexia (General disorders) | 54 (62) | 56 (80)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 6 (6) | 5 (5)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 37 (37) | 39 (39)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 2 (4)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 20 (24)
Vaccination site induration (General disorders) | 2 (2) | 4 (4)
Vaccination site swelling (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (33) | 30 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT02907216/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02907216/SAP_001.pdf